CLINICAL TRIAL: NCT03085069
Title: An Open-label, Single-arm, Multi-center, Phase 2 Study to Evaluate SHR-1210(Anti-PD-1 Antibody) in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate SHR-1210 in Patients With Advanced or Metastatic NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-II-201-NSCLC
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms Nec; Lung Disease; Respiratory Tract Disease; Neoplasm, Bronchial; Carcinoma, Bronchogenic
Keywords: PD-1; PD-L1; SHR-1210
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Respiratory Tract Diseases; Bronchial Neoplasms; Carcinoma, Bronchogenic | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PD-L1 expression in tumor ≥ 50% (Experimental): Subjects receive SHR-1210 intravenous at the dose 200mg on Day 1 every 2 weeks
  Interventions: Biological: SHR-1210
- PD-L1 expression in tumor ≥25-50% (Experimental): Subjects receive SHR-1210 intravenous at the dose 200mg on Day 1 every 2 weeks
  Interventions: Biological: SHR-1210
- PD-L1 expression in tumor ≥ 1-25% (Experimental): Subjects receive SHR-1210 intravenous at the dose 200mg on Day 1 every 2 weeks
  Interventions: Biological: SHR-1210
- PD-L1 expression in tumor < 1% (Experimental): Subjects receive SHR-1210 intravenous at the dose 200mg on Day 1 every 2 weeks
  Interventions: Biological: SHR-1210

INTERVENTIONS:
Biological: SHR-1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody

SUMMARY:
This is an open-label, single-arm, multi-center, phase 2 Study to evaluate SHR-1210(anti-PD-1 antibody) in in adult Chinese patients with advanced or metastatic non-small cell lung cancer who failed or progressed to prior first-line systemic treatment.

Enrolled subjects will be assigned to 4 cohorts on the basis of PD-L1 expression in tumor cells(<1%, ≥1%-25%, ≥25%-50%, ≥50%) all will be treated with the standard SHR-1210 dose (200mg) , Q2W, until documented progressive disease (PD) occurs. Subjects will return to the clinic once every two weeks. Radiographic disease assessments will be performed every 6 weeks.

The primary study hypothesis is that treatment with SHR-1210 improves Objective Response Rate when compare with standard second-line therapy, no matter how much PD-L1 expression in tumor.

DETAILED DESCRIPTION:
In similar clinical trials, anti-PD-1 and anti-PD-L1 antibodies produce durable responses in approximately 20% of unselected patients with advanced non-small-cell lung cancer. Developing reliable, validated biomarkers that identify patients with an increased probability of response to these antibodies remains a challenge.

Because the PD-1 pathway may be a key mechanism of immune escape in a subgroup of patients with non-small-cell lung cancer, PD-L1 expression in tumor or inflammatory cells is a candidate biomarker. However, PD-L1 expression has not been formally validated as a biomarker in contemporaneously collected tumor tissue.

Additionally the purpose of the study is to assess the correlation between the expression of PD-L1 in the tumor and the response to treatment with SHR-1210 in non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically- or cytologically- documented NSCLC who present with Stage IIIB-IV disease (according to version 7 of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology), or disease recurrence or progression following multi-modal therapy (radiation therapy, surgical resection or radical chemo-radiotherapy in locally advanced disease).
2. Fresh cutting specimens or hollow needle aspiration specimens must be provided. A formalin fixed, paraffin-embedded (FFPE) tumor tissue block or unstained slides of tumor sample (must be recent) must be available for biomarker evaluation. In the case of unstained slides, a minimum of 8 slides are necessary to conduct the planned biomarker analyses. Specimens must be received by the central lab prior to randomization. Biopsy should be excisional, incisional or core needle.
3. Subjects must have experienced disease recurrence or progression during or after one prior platinum-containing doublet chemotherapy regimen for advanced or metastatic disease:

   1. Subjects who received maintenance therapy (non-progressors with platinum-based doublet chemotherapy) and progressed are eligible.
   2. Subjects who received adjuvant or neoadjuvant platinum-doublet chemotherapy (after surgery and/or radiation therapy) and developed recurrent or metastatic disease within 6 months of completing therapy are eligible.
   3. Subjects with recurrent disease > 6 months after adjuvant or neoadjuvant platinum based chemotherapy, who also subsequently progressed during or after a platinum-doublet regimen given to treat the recurrence, are eligible.
4. Subjects with sensitizing EGFR mutation positive or ALK rearrangement positive, must have experienced disease recurrence or progression during or after one prior tyrosine kinase inhibitor regimen, who also have PD-L1 expression in tumor ≥ 50%, are eligible.
5. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria; Radiographic Tumor Assessment performed within 28 days of randomization.
6. Eastern Cooperative Oncology Arm (ECOG) performance status of ≤ 1.
7. All baseline laboratory requirements will be assessed and should be obtained within -14 days of randomization. Screening laboratory values must meet the following criteria.

   1. Absolute neutrophil count ≥ 1.5 × 109/L (1500/mm3)
   2. Platelets ≥ 80× 109/L (100,000/mm3)
   3. Hemoglobin ≥ 9.0 g/dL (90 g/L)
   4. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal(ULN); for subjects with liver metastases, ALT and AST ≤ 5 × ULN
   6. Serum creatinine ≤1.5 × ULN or creatinine clearance > 45 mL/minute (using Cockcroft/Gault formula)
8. Female participants of childbearing potential must have a negative serum pregnancy test within -7 days of randomization and must be willing to use very efficient barrier methods of contraception or a barrier method plus a hormonal method starting with the screening visit through 60 days (about 5 drug half-life + menstrual cycle) after the last dose of SHR-1210. Male participants with a female partner(s) of child-bearing potential must be willing to use very efficient barrier methods of contraception from screening through 120 days (about 5 drug half-life + sperm depletion cycle) after the last dose of SHR-1210.
9. Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests including completion of patient reported outcomes questionnaires and other requirements of the study. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.

Exclusion Criteria:

1. Target Disease Exceptions

   1. Subjects with active CNS metastases are excluded. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
   2. Subjects with carcinomatous meningitis.
2. Medical History and Concurrent Diseases

   1. Subjects with active, known or suspected autoimmune disease. Subjects in conditions not expected to recur in the absence of an external trigger are permitted to enroll.
   2. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
   3. Prior therapy with immunostimulatory medications or tumor vaccines within 6 months.
   4. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
   5. Treatment with any investigational agent within 5 half-life of the agent, before the first administration of study treatment.
   6. Subjects with a history of interstitial lung disease.
   7. Subjects received lung radiation therapy within 6 months.
   8. Other active malignancy requiring concurrent intervention.
   9. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, endometrial, cervical/dysplasia) are excluded unless a complete remission was achieved at least 5 years prior to study entry.
   10. Subjects have had prior chemotherapy within 3 weeks prior to study, or have had prior targeted small molecule therapy within 1 weeks prior to study, or have had prior radiation therapy or surgical operation within 4 weeks prior to study, or have had prior anti-tumor biotherapy within 3 weeks prior to study. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug.
   11. Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment
   12. Subjects with active pulmonary tuberculosis.
   13. Subjects with hemoptysis or hemorrhagic quantity per day is 2.5 ml or above within 4 weeks prior to study.
3. Physical and Laboratory Test Findings

   1. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
   2. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. (HBV: HBsAg positive and HBV DNA ≥ 500 IU/mL ; HVC: HCV RNA positive and abnormal liver function).
4. Allergies and Adverse Drug Reaction

   1. History of severe hypersensitivity reactions to other monoclonal antibodies.
   2. History of severe hypersensitivity reaction to intravenous infusion.
5. Other Exclusion Criteria Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2023-08-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Determined using RECIST v1.1 criteria, up to approximately 1 year
  Objective response is defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.

SECONDARY OUTCOMES:
Duration of Response Rate | Determined using RECIST v1.1 criteria, up to approximately 1 year
Overall Survival Rate at 12-month | up to approximately 1 year
Progression-Free Survival | Determined using RECIST v1.1 criteria, up to approximately 1 year
Number of participants with treatment-related adverse events (AEs) | up to approximately 1 year
  assessed by NCI-CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Wei Shi, MD, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (1):
- Guangdong Lung Cancer Institute (GLCI),Guangdong General Hospital (GGH), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang JJ, Huang C, Fan Y, Pan H, Feng J, Jiang L, Li XY, Liu XQ, Xiong JP, Zhao YQ, Cheng Y, Ma R, Wang J, Wang Y, Liu YH, Lin DM, Wang T, Shi W, Zou J, Wu YL. Camrelizumab in different PD-L1 expression cohorts of pre-treated advanced or metastatic non-small cell lung cancer: a phase II study. Cancer Immunol Immunother. 2022 Jun;71(6):1393-1402. doi: 10.1007/s00262-021-03091-3. Epub 2021 Oct 20. PMID 34668977